CLINICAL TRIAL: NCT07333716
Title: Efficacy and Safety of Desloratadine as Adjuvant Therapy in Patients With Ulcerative Colitis
Brief Title: Desloratadine in Patients With Ulcerative Colitis
Acronym: UC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Romisaa Raafat Abd Alnapy Mohamed, clinical pharmacy resident, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/2025 TRop1
Record Dates: First submitted 2026-01-01; First posted 2026-01-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis (UC); Ulcerative Colitis
Keywords: Ulcerative Colitis; Desloratadine
MeSH Terms: conditions — Colitis, Ulcerative | interventions — desloratadine; Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Control group) (Placebo Comparator): which will receive mesalamine (standard treatment ) 1000 mg three times daily for 3 months and serve as the control group
  Interventions: Drug: mesalamine
- Group II (Desloratadine group) (Active Comparator): which will receive mesalamine (standard treatment )1000 mg three times daily plus desloratadine 5 mg once daily for 3 months
  Interventions: Drug: Desloratadine

INTERVENTIONS:
Drug: Desloratadine — mesalamine 1000 mg three times daily plus desloratadine 5 mg once daily for 3 months.
  Arms: Group II (Desloratadine group)
Drug: mesalamine — mesalamine 1000 mg three times daily for 3 months
  Arms: Group I (Control group)

SUMMARY:
The purpose of this study is to investigate safety and therapeutic efficacy of antihistamine (desloratadine) on inflammation and disease activity when administered as adjuvant therapies with the traditional therapy 5-aminosalisylic acid (mesalamine) in patients with mild to moderate ulcerative colitis.

DETAILED DESCRIPTION:
Ulcerative colitis is a chronic inflammatory autoimmune disease affecting the colon. The World Health Organization has classified it as a relatively new treatment-resistant disease, and its prevalence has reportedly increased significantly in Egypt. A preclinical study was conducted to evaluate desloratadine as a potential therapeutic agent for ulcerative colitis, based on its known anti-inflammatory and antioxidant properties. The study concluded that desloratadine effectively alleviated experimental ulcerative colitis. This positive effect is attributed to its anti-inflammatory and antioxidant properties, which work by regulating mast cell activity and inhibiting histamine release.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female sex.
* patients with age ranged from 18 to 65.
* patients with active mild and moderate ulcerative colitis according to American College of Gastroenterology (ACG) Clinical Guideline.
* Patients treated with 5-aminosalisylic acid (mesalamine).

Exclusion Criteria:

* Patients with severe UC
* Significant liver or kidney function abnormalities
* Pregnant or lactating females
* Treatment with systemic or rectal steroids
* Treatment with immunosuppressant or biological therapies
* Known allergy to desloratadine or any ingredient in the formulation
* Patients with other inflammatory diseases
* Patients with history of colon cancer
* Patients with complete or partial colectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in disease activity and severity | over a 3 month follow -up period
  Change in disease activity and severity through Partial Mayo Scoring Index (PMSI) and Truelove and Witt's classification

SECONDARY OUTCOMES:
Change in serum biomarkers | Change from baseline in serum biomarker over 3 months
  Change in serum biomarkers of inflammation and oxidative stress (TNF-α & MDA)

CONTACTS AND LOCATIONS:
Overall Officials: Romisaa R Abd Alnapy, Principal Investigator — Tanta University
Locations (1):
- Menofia university Hospitals, Shibīn al Kawm, Menofia, Egypt

IPD SHARING:
Plan to Share IPD: No